CLINICAL TRIAL: NCT01405534
Title: Evaluation of the Occurrence of Acute Complications Caused by a Central Venous Catheter Placement: Observational, Prospective, Monocentric Study
Brief Title: Evaluation of the Occurrence of Acute Complications Caused by a Central Venous Catheter Placement
Acronym: VVC
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: VVC
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Anesthesia
Keywords: Catheterization, Central Venous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Central venous catheter: All patients who require the placement of a central venous catheter

SUMMARY:
It is an observational, prospective, monocentric study. The purpose of the study is to assess the acute complications rate caused by a central venous catheter placement.

All the patients who require a central venous placement could be enrolled in the study.

The study will not change the usual practice. The placement will be on day 1 and patients will be contacted by phone on day 7 to identify potential complications and to assess pain.

Anaesthesia staff will keep patients under surveillance to control the absence of late complications.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18.
* Patient who requires the placement of a central venous catheter (a portacath (PAC), a peripherally inserted central catheter (PICC) or a tunnelled catheter).
* Patient able to understand, read and write French.
* Mandatory affiliation with a health insurance system.

Exclusion Criteria:

* Active infection at placement of the central venous catheter.
* Patient who can't be contacted by phone.
* Patient who is likely to have a femoral venous catheter placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patient who require the placement of a central venous catheter
Sampling Method: Non-Probability Sample
Enrollment: 1780 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Estimate the acute complications rate | From day 1 to day 7
  Placement of the central venous catheter on day 1 and follow-up of potential acute complications

SECONDARY OUTCOMES:
Assess the preoperative anxiety | On day 1
  By means of Beck anxiety inventory
Assess patients satisfaction about the catheter | On day 7
  By means of a questionnary filled in by patients at home
Assess postoperative pain | On day 1 and on day 7
  The pain will be assessed on day 1 by a visual analogic scale and on day 7 by a verbal numeric scale
Assess the rate of late complications | Up to 1 year
  The anaesthesia staff will keep patients under surveillance for potential late complications.

CONTACTS AND LOCATIONS:
Overall Officials: Hervé ROSAY, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France

REFERENCES:
- [Background] Gambotti L, Perol D, Frering B, Kaemmerlen P, Coronel B, Sebban H, Bulso V, Bachelot V, Chauvin F, Bachmann P. Safety of percutaneous internal jugular catheterization in cancer patients: prospective observational study. J Vasc Access. 2004 Oct-Dec;5(4):161-7. doi: 10.1177/112972980400500405. PMID 16596560
- [Background] Maki DG, Kluger DM, Crnich CJ. The risk of bloodstream infection in adults with different intravascular devices: a systematic review of 200 published prospective studies. Mayo Clin Proc. 2006 Sep;81(9):1159-71. doi: 10.4065/81.9.1159. PMID 16970212
- [Background] Burns KE, McLaren A. Catheter-related right atrial thrombus and pulmonary embolism: a case report and systematic review of the literature. Can Respir J. 2009 Sep-Oct;16(5):163-5. doi: 10.1155/2009/751507. PMID 19851535
- [Background] Kim HJ, Yun J, Kim HJ, Kim KH, Kim SH, Lee SC, Bae SB, Kim CK, Lee NS, Lee KT, Park SK, Won JH, Park HS, Hong DS. Safety and effectiveness of central venous catheterization in patients with cancer: prospective observational study. J Korean Med Sci. 2010 Dec;25(12):1748-53. doi: 10.3346/jkms.2010.25.12.1748. Epub 2010 Nov 24. PMID 21165289
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: central line-associated blood stream infections--United States, 2001, 2008, and 2009. MMWR Morb Mortal Wkly Rep. 2011 Mar 4;60(8):243-8. PMID 21368740
- [Background] Yacopetti N, Alexandrou E, Spencer TR, Frost SA, Davidson PM, O'Sullivan G, Hillman KM. Central venous catheter insertion by a clinical nurse consultant or anaesthetic medical staff: a single-centre observational study. Crit Care Resusc. 2010 Jun;12(2):90-5. PMID 20513216